CLINICAL TRIAL: NCT06483191
Title: Acceptability and Feasibility of Acceptance and Commitment Therapy in Total Knee Arthroplasty Patients
Brief Title: IMProving Outcomes With ACT After Knee Surgery
Acronym: IMPACTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); Trauma and Orthopaedics Research Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23007RN-SW
Record Dates: First submitted 2024-01-31; First posted 2024-07-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: A single centred, parallel group, randomised controlled trial
Who Masked: Investigator
Masking Description: The Chief Investigator will be blinded to what group patients are randomised to. It will not be possible to blind the patients, research team or physiotherapists involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Patients will attend a half-day virtual pre-operative ACT group workshop delivered by physiotherapists. Intervention group patients will also receive booster post-operative ACT text messages once a week for 6 weeks and a telephone follow-up with a physiotherapist at 6-8 weeks. The workshop, text messages and follow-up with a physiotherapist will be in addition to standard care.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control (No Intervention): Patients in the control group will receive standard care; All patients should attend a 1-hour face-to-face group pre-operative education class. Patients in either group will have access to a helpline where they can speak to a nurse to discuss any problems or concerns. All patients will also receive a follow-up phone call from a nurse within 5 days of discharge to check their progress and will attend a 6-12 week follow-up clinic with their surgeon.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — A half-day pre-operative virtual ACT group workshop, booster post-operative ACT text messages once a week for 6 weeks and a telephone follow-up with a physiotherapist at 6-8 weeks (all in addition to standard care).
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy (ACT)

SUMMARY:
Regarding psychosocial factors and outcomes in total knee arthroplasty (TKA), most of the current literature and the investigators' previous work suggest that depression, anxiety and pre-operative pain strongly predict worse outcomes following TKA. Despite some conflicting evidence, on the whole, the current literature suggests that psychological intervention in TKA patients could help to improve outcomes. In recent years, Acceptance and Commitment Therapy (ACT) has been receiving more attention as it may be more effective than the more traditional cognitive behavioural therapy in treating older people with chronic pain. ACT includes a combination of acceptance and mindfulness methods along with activation and behaviour change methods.

There have been several studies examining ACT in patients undergoing orthopaedic surgery. These studies have found that attending a pre-operative ACT workshop and receiving text messages reinforcing ACT can reduce use of pain medication, reduce post-operative pain and improve function following surgery. There are also two study protocols published which plan to investigate ACT in TKA patients but the findings of these studies are yet to be reported.

In this feasibility study, the investigators propose to investigate the acceptability and feasibility of a pre-operative ACT workshop in TKA patients considered to be at risk of poorer outcome based on a depression score. If found to be acceptable and feasible to both patients and those who will deliver the ACT sessions, a larger study will be performed.

DETAILED DESCRIPTION:
Regarding psychosocial factors and outcomes in total knee arthroplasty (TKA), most of the current literature suggests that depression, anxiety and pre-operative pain strongly predict worse outcomes following TKA. The investigators' previous work agreed with these findings and other psychological factors, such as neuroticism, pain catastrophising and self-blame were associated with worse outcomes up to 1 year following TKA whilst conscientiousness, pain self-efficacy and extraversion were associated with better outcomes up to 1 year following TKA. These psychological factors have been less consistently associated with outcomes following joint arthroplasty in other papers and several papers have found no evidence or conflicting evidence that depression or anxiety are associated with outcomes following TKA. Despite some conflicting evidence, on the whole, the current literature suggests that psychological intervention in TKA patients could help to improve outcomes.

To date, few studies have randomised patients to a psychological intervention or control group to determine whether intervention could improve outcomes following TKA or total hip arthroplasty (THA). A systematic review by Bay et al. (2018) reported that the current literature, which is still in its infancy, does not support routine psychological interventions for TKA or THA. This review included seven studies of randomised controlled trials (RCTs) of psychological interventions which involved active patient participation measured with patient reported outcomes in THA or TKA patients. Only two of these studies found psychological interventions to be effective in improving at least one patient reported outcome. One study used a combination of cognitive behaviour therapy and relaxation therapy in THA patients and this was found to significantly improve hip function at 1-year follow-up. In the second study, guided imagery improved gait velocity 6 months after TKA, and reduced knee pain 3 weeks after surgery compared to the control group.

Recently, ACT has been receiving more attention as it may be more effective than the more traditional cognitive behavioural therapy in treating older people with chronic pain. ACT includes a combination of acceptance and mindfulness methods along with activation and behaviour change methods. The goal of ACT is to enhance psychological and behavioural flexibility by cultivating the six inter-rated skills of acceptance, cognitive defusion, present-moment awareness, values clarification, committed action, and perspective taking.

In the current literature, there have been several studies examining ACT in patients undergoing orthopaedic surgery. One study included 88 veterans who were undergoing orthopaedic surgery (including TKA, THA, shoulder and spine). Half of the patients were randomised to standard care and the other half attended a 1-day ACT workshop pre-operatively in addition to standard care. Pain levels and opioid use were assessed up to 3 months following surgery. The intervention group achieved pain and opioid cessation sooner than those in the control group. Increases in pain acceptance and values-based behaviour, processes targeted in ACT, were related to better outcomes. The other study included 76 patients who underwent operative fixation of a traumatic upper or lower extremity fracture. Patients were randomised to the intervention group, who received twice-daily text messages communicating an ACT-based intervention for the first 2 weeks after surgery, or the control group, who received no text messages. At baseline, patients completed paper forms comprising a basic demographics questionnaire and baseline patient-reported outcomes. Two weeks following surgery, patients again completed the patient reported outcomes and had an opioid medication pill count. On average, the intervention group used 36.5% fewer opioid tablets compared to the control group (intervention group average: 26.1 (SD 21.4) tablets, control group average: 41.1 (SD 22.0) tablets). The intervention group also reported significantly lower post-operative pain compared to the control group. The same group of authors then investigated ACT using the same intervention (text messages sent twice a day for 2 weeks) to a total of 45 THA and TKA patients who had their surgeries delayed due to the Covid-19 pandemic. They found that the ACT group showed improved function and slowed decline compared to the other 45 in the control group who did not receive any text messages.

There are also two study protocols published which plan to investigate ACT in TKA patients but the findings of these studies are yet to be reported.

Based on the investigators' previous work, psychological factors are associated with TKA outcomes, therefore, in this feasibility study, the investigators propose to examine the acceptability and feasibility of a pre-operative ACT workshop in TKA patients considered to be at risk of poorer outcomes based on a depression score. If found to be acceptable and feasible to both patients and those who will deliver the ACT sessions, a larger study will be performed to determine whether ACT can improve outcomes in TKA patients.

The aim of this feasibility study is to determine the acceptability and feasibility of a half day pre-operative ACT workshop, ACT text messages and follow-up with a physiotherapist in a cohort of patients undergoing TKA who have been identified as having a higher likelihood of a below average post-operative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old scheduled for routine primary elective TKA.
* Participants must have a functional level of spoken and written English and be able to complete the online pre-operative psychosocial questionnaire independently.
* Patients must have scored 10 or more on the Depression subscale of the (Depression, Anxiety and Stress Scale) DASS-21 of the pre-operative psychosocial questionnaire.

Exclusion Criteria:

* Any patient who does not have access to a mobile phone to receive the booster text messages, or online facilities to answer online questionnaires.
* Any patient who has a significant change (≥3 months) in scheduled date of surgery i.e. has a delayed surgery or surgery earlier than expected.
* Any patient who does not attend the pre-operative education class.
* Any patient scheduled for revision, uni-compartmental or bilateral TKA.
* Any patient who has further orthopaedic surgery planned in the next 3 months.
* Any patient who cannot commit to the schedule of events.
* Any patient currently receiving any other "talking therapy".

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability and feasibility of the intervention | 6-8 weeks
  Acceptability of the intervention will be assessed via an online questionnaire to be completed by patients who were randomised to the intervention group. Patients in the control group will also complete a modified set of questions to determine how they felt being randomised to the standard care group and whether they would have liked more support.

SECONDARY OUTCOMES:
Change in Oxford Knee Score (OKS) from pre-operation to 3 months | Preoperation, 3 months
  The OKS will be completed by participants online, with a score ranging from 0 (worst score possible) - 48 (best score possible).
EuroQol-5D-5L | Pre-operation, 3 months
  The EQ-5D-5L will be completed by participants online. A single score will be derived which ranges from -0.594 to 1, where 0 is death and 1 is full health.
EuroQoL-5D Visual Analogue Scale (VAS) | Pre-operation, 3 months
  The EQ-5D VAS will also be scored from 0 (worst health possible) - 100 (best health possible).
Pain Interference | Pre-operation, 3 months
  Pain interference will be completed by all patients recruited to the study (following consent and prior to randomisation before attending the pre-operative ACT workshop for the intervention group) and at 3 months post-operatively.
Acceptance and Action Questionnaire (AAQ) | Pre-operation, 3 months
  The Acceptance and Action Questionnaire (AAQ) will be completed by all patients recruited to the study (following consent and prior to randomisation before attending the pre-operative ACT workshop for the intervention group) and at 3 months post-operatively.
Chronic Pain Acceptance Questionnaire-2 (CPAQ-2) | Pre-operation, 3 months
  The Chronic Pain Acceptance Questionnaire-2 (CPAQ-2) will be completed by all patients recruited to the study (following consent and prior to randomisation before attending the pre-operative ACT workshop for the intervention group) and at 3 months post-operatively.
Chronic Pain Values Inventory (CPVI) | Pre-operation, 3 months
  The Chronic Pain Values Inventory (CPVI) will be completed by all patients recruited to the study (following consent and prior to randomisation before attending the pre-operative ACT workshop for the intervention group) and at 3 months post-operatively.
Length of hospital stay | 3 months
  Total length of hospital stay will be calculated using date of discharge and date of operation.
Post-discharge Non-Scheduled Contact | 3 months
  This will include inpatient or outpatient physiotherapy sessions, unscheduled face-to-face contact with nurse, orthopaedic surgeon or physiotherapist, phone calls to physiotherapist team, helpline calls, out of hours attendances, A&E attendances, hospital readmissions and returns to theatre up to 90 days post-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Napier, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Musgrave Park Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorel JC, Veltman ES, Honig A, Poolman RW. The influence of preoperative psychological distress on pain and function after total knee arthroplasty: a systematic review and meta-analysis. Bone Joint J. 2019 Jan;101-B(1):7-14. doi: 10.1302/0301-620X.101B1.BJJ-2018-0672.R1. PMID 30601044
- [Background] Hernandez C, Diaz-Heredia J, Berraquero ML, Crespo P, Loza E, Ruiz Iban MA. Pre-operative Predictive Factors of Post-operative Pain in Patients With Hip or Knee Arthroplasty: A Systematic Review. Reumatol Clin. 2015 Nov-Dec;11(6):361-80. doi: 10.1016/j.reuma.2014.12.008. Epub 2015 Apr 1. English, Spanish. PMID 25840826
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] Alattas SA, Smith T, Bhatti M, Wilson-Nunn D, Donell S. Greater pre-operative anxiety, pain and poorer function predict a worse outcome of a total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3403-3410. doi: 10.1007/s00167-016-4314-8. Epub 2016 Oct 12. PMID 27734110
- [Background] Lungu E, Vendittoli PA, Desmeules F. Preoperative Determinants of Patient-reported Pain and Physical Function Levels Following Total Knee Arthroplasty: A Systematic Review. Open Orthop J. 2016 Jun 23;10:213-31. doi: 10.2174/1874325001610010213. eCollection 2016. PMID 27398109
- [Background] Hofstede SN, Gademan MG, Vliet Vlieland TP, Nelissen RG, Marang-van de Mheen PJ. Preoperative predictors for outcomes after total hip replacement in patients with osteoarthritis: a systematic review. BMC Musculoskelet Disord. 2016 May 17;17:212. doi: 10.1186/s12891-016-1070-3. PMID 27184266
- [Background] Lindner M, Nosseir O, Keller-Pliessnig A, Teigelack P, Teufel M, Tagay S. Psychosocial predictors for outcome after total joint arthroplasty: a prospective comparison of hip and knee arthroplasty. BMC Musculoskelet Disord. 2018 May 22;19(1):159. doi: 10.1186/s12891-018-2058-y. PMID 29788969
- [Background] Belford K, Gallagher N, Dempster M, Wolfenden M, Hill J, Blaney J, O'Brien S, Smit AM, Botha P, Molloy D, Beverland D. Psychosocial predictors of outcomes up to one year following total knee arthroplasty. Knee. 2020 Jun;27(3):1028-1034. doi: 10.1016/j.knee.2020.03.006. Epub 2020 Apr 13. PMID 32299757
- [Background] Vissers MM, Bussmann JB, Verhaar JA, Busschbach JJ, Bierma-Zeinstra SM, Reijman M. Psychological factors affecting the outcome of total hip and knee arthroplasty: a systematic review. Semin Arthritis Rheum. 2012 Feb;41(4):576-88. doi: 10.1016/j.semarthrit.2011.07.003. Epub 2011 Oct 28. PMID 22035624
- [Background] Magklara E, Burton CR, Morrison V. Does self-efficacy influence recovery and well-being in osteoarthritis patients undergoing joint replacement? A systematic review. Clin Rehabil. 2014 Sep;28(9):835-46. doi: 10.1177/0269215514527843. Epub 2014 Mar 25. PMID 24668361
- [Background] Burns LC, Ritvo SE, Ferguson MK, Clarke H, Seltzer Z, Katz J. Pain catastrophizing as a risk factor for chronic pain after total knee arthroplasty: a systematic review. J Pain Res. 2015 Jan 5;8:21-32. doi: 10.2147/JPR.S64730. eCollection 2015. PMID 25609995
- [Background] Riddle DL, Wade JB, Jiranek WA, Kong X. Preoperative pain catastrophizing predicts pain outcome after knee arthroplasty. Clin Orthop Relat Res. 2010 Mar;468(3):798-806. doi: 10.1007/s11999-009-0963-y. Epub 2009 Jul 8. PMID 19585177
- [Background] Riddle DL, Jensen MP, Ang D, Slover J, Perera R, Dumenci L. Do Pain Coping and Pain Beliefs Associate With Outcome Measures Before Knee Arthroplasty in Patients Who Catastrophize About Pain? A Cross-sectional Analysis From a Randomized Clinical Trial. Clin Orthop Relat Res. 2018 Apr;476(4):778-786. doi: 10.1007/s11999.0000000000000001. PMID 29543659
- [Background] Bletterman AN, de Geest-Vrolijk ME, Vriezekolk JE, Nijhuis-van der Sanden MW, van Meeteren NL, Hoogeboom TJ. Preoperative psychosocial factors predicting patient's functional recovery after total knee or total hip arthroplasty: a systematic review. Clin Rehabil. 2018 Apr;32(4):512-525. doi: 10.1177/0269215517730669. Epub 2017 Sep 19. PMID 28922942
- [Background] Khatib Y, Madan A, Naylor JM, Harris IA. Do Psychological Factors Predict Poor Outcome in Patients Undergoing TKA? A Systematic Review. Clin Orthop Relat Res. 2015 Aug;473(8):2630-8. doi: 10.1007/s11999-015-4234-9. Epub 2015 Mar 20. PMID 25791440
- [Background] Bay S, Kuster L, McLean N, Byrnes M, Kuster MS. A systematic review of psychological interventions in total hip and knee arthroplasty. BMC Musculoskelet Disord. 2018 Jun 21;19(1):201. doi: 10.1186/s12891-018-2121-8. PMID 30037341
- [Background] Berge DJ, Dolin SJ, Williams AC, Harman R. Pre-operative and post-operative effect of a pain management programme prior to total hip replacement: a randomized controlled trial. Pain. 2004 Jul;110(1-2):33-9. doi: 10.1016/j.pain.2004.03.002. PMID 15275749
- [Background] Jacobson AF, Umberger WA, Palmieri PA, Alexander TS, Myerscough RP, Draucker CB, Steudte-Schmiedgen S, Kirschbaum C. Guided Imagery for Total Knee Replacement: A Randomized, Placebo-Controlled Pilot Study. J Altern Complement Med. 2016 Jul;22(7):563-75. doi: 10.1089/acm.2016.0038. Epub 2016 May 23. PMID 27214055
- [Background] Wetherell JL, Petkus AJ, Alonso-Fernandez M, Bower ES, Steiner AR, Afari N. Age moderates response to acceptance and commitment therapy vs. cognitive behavioral therapy for chronic pain. Int J Geriatr Psychiatry. 2016 Mar;31(3):302-8. doi: 10.1002/gps.4330. Epub 2015 Jul 28. PMID 26216753
- [Background] McCracken LM, Vowles KE. Acceptance and commitment therapy and mindfulness for chronic pain: model, process, and progress. Am Psychol. 2014 Feb-Mar;69(2):178-87. doi: 10.1037/a0035623. PMID 24547803
- [Background] Roddy MK, Boykin DM, Hadlandsmyth K, Marchman JN, Green DM, Buckwalter JA 4th, Garvin L, Zimmerman B, Bae J, Cortesi J, Rodrigues M, Embree J, Rakel BA, Dindo L. One-day Acceptance and Commitment Therapy workshop for preventing persistent post-surgical pain and dysfunction in at-risk veterans: A randomized controlled trial protocol. J Psychosom Res. 2020 Nov;138:110250. doi: 10.1016/j.jpsychores.2020.110250. Epub 2020 Sep 15. PMID 32961500
- [Background] Dindo L, Zimmerman MB, Hadlandsmyth K, StMarie B, Embree J, Marchman J, Tripp-Reimer T, Rakel B. Acceptance and Commitment Therapy for Prevention of Chronic Postsurgical Pain and Opioid Use in At-Risk Veterans: A Pilot Randomized Controlled Study. J Pain. 2018 Oct;19(10):1211-1221. doi: 10.1016/j.jpain.2018.04.016. Epub 2018 May 17. PMID 29777950
- [Background] Anthony CA, Rojas EO, Keffala V, Glass NA, Shah AS, Miller BJ, Hogue M, Willey MC, Karam M, Marsh JL. Acceptance and Commitment Therapy Delivered via a Mobile Phone Messaging Robot to Decrease Postoperative Opioid Use in Patients With Orthopedic Trauma: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 29;22(7):e17750. doi: 10.2196/17750. PMID 32723723
- [Background] March MK, Harmer A, Godfrey E, Venkatesh S, Thomas B, Dennis S. The KOMPACT-P study: Knee Osteoarthritis Management with Physiotherapy informed by Acceptance and Commitment Therapy-Pilot study protocol. BMJ Open. 2020 Jun 3;10(6):e032675. doi: 10.1136/bmjopen-2019-032675. PMID 32499254